CLINICAL TRIAL: NCT03899922
Title: Monitoring Drug-induced Uveitis
Acronym: UVETOX
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-19-07
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Uveitis; Uveitis Drug-Induced; Eye Diseases; Uvea--Diseases
Keywords: Uvea toxicity; chemotherapies; drugs
MeSH Terms: conditions — Uveitis; Eye Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Uveitis induced by drugs and chemotherapies: Case reported in the World Health Organization (WHO) of uveitis of patient treated by a drug, with a chronology compatible with the drug toxicity
  Interventions: Drug: Drugs inducing uveitis

INTERVENTIONS:
Drug: Drugs inducing uveitis — Drugs susceptible to induce uveitis

SUMMARY:
Several drugs and chemotherapies seem to induce uveitis. This study investigates reports of uveitis, including the International classification of disease ICD-10 for treatments in the World Health Organization (WHO) global Individual Case Safety Report (ICSR) database (VigiBase).

DETAILED DESCRIPTION:
Several drugs and chemotherapies seem to have an impact on the eyes and are responsible of uveitis. Those are poorly described, due to the modification of the pharmacopeia, and the recent recognition of several of these adverse events. This study investigates the main characteristics of patients affected by uveitis side effect imputed to drugs. A causality assessment according to the WHO-UMC (World Health Organization - Uppsala Monitoring Center) is systematically applied.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the WHO's pharmacovigilance database till 01/04/2019

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a drug that could be reported in the WHO's pharmacovigilance database
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Eye toxicities of drugs Identification and report of cases of uevitis associated with drugs | to 01/04/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports

SECONDARY OUTCOMES:
Causality assessment of reported uveitis according to the WHO system | to 01/04/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
All relevants statisticals associations between type of uveitis and the category of drug | to 01/04/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
All relevants statisticals associations between other concomittants immune related adverse events and uveitis induced by drugs | to 01/04/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Duration of treatment when uveitis happen (role of cumulative dose) | to 01/04/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
All relevants statisticals associations between drug-drug interactions and adverse events | to 01/04/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
All relevants statisticals associations between pathologies (cancer) for which the incriminated drugs have been prescribed, and occurence of uveitis | to 01/04/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
All relevants statisticals associations between characteristics of the population and occurence of uveitis adverse event | to 01/04/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided